CLINICAL TRIAL: NCT01409642
Title: Pilot Feasibility Trial of Positive Family Interaction Therapy
Brief Title: Family Focused Treatment of Pediatric Obsessive Compulsive Disorder
Acronym: PFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Tara Peris, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K23MH085058 (NIH)
Record Dates: First submitted 2010-10-12; First posted 2011-08-04 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individual Child CBT (Active Comparator): 12 sessions of individual child-focused cognitive behavior therapy with a parent component
  Interventions: Behavioral: Individual Child CBT
- Positive Family Interaction Therapy (Experimental): 12 sessions of standard individual child CBT plus six sessions of positive family interaction therapy (PFIT)
  Interventions: Behavioral: Positive Family Interaction Therapy

INTERVENTIONS:
Behavioral: Individual Child CBT — 12 sessions of individual child focused cognitive behavior therapy with a parent component
  Other Names: child cognitive behavior therapy
  Arms: Individual Child CBT
Behavioral: Positive Family Interaction Therapy — Six sessions of family-focused treatment for childhood OCD administered as an adjunct to 12 sessions of child CBT
  Arms: Positive Family Interaction Therapy
Behavioral: Positive Family Interaction Therapy — Positive Family Interaction Therapy (PFIT) is a 6-session treatment designed to be used as an adjunct to standard child CBT in cases where OCD is complicated by challenging family dynamics.
  Other Names: PFIT
  Arms: Positive Family Interaction Therapy

SUMMARY:
Pediatric obsessive compulsive disorder (OCD) is a chronic, impairing condition that accrues significant concurrent and long-term risk to affected youth (Piacentini et al. 2003; Pine et al. 1998). Although a host of pharmacological and psychosocial treatments have proliferated over the past decade (Barrett et al., 2008), many youth fail torespond to treatment and many who do respond continue to exhibit lingering symptoms and impairment. Thus, there is still much to be done by way of optimizing treatment outcomes for pediatric OCD.

Increasingly, efforts to improve existing treatments have focused on aspects of the family environment that may affect treatment adherence and the maintenance of therapeutic gains. Such work suggests that parental accommodation and criticism are common characteristics of the home environment for both adults and children with OCD (Calvocoressi et al., 1999; Peris, Roblek, Langley, Chang, McCracken, & Piacentini, 2008; Van Noppen et al., 1991) and that, in adult samples, these family features are associated with poorer treatment outcome and greater risk of relapse (Amir, Freshman, & Foa, 2000; Chambless & Steketee, 1999;Leonard et al., 1993). These family-level variables are logical targets for intervention, particularly among treatment refractory groups of youth with OCD. However, they often are unaddressed in extant interventions.

The current study tests a novel intervention that specifically targets family accommodation and conflict in an effort to foster an environment that supports a graded exposure approach to treatment. The proposed treatment, Positive Family Interaction Therapy (PFIT), is composed of an innovative blend of techniques that address several potential barriers to treatment. First, the treatment is guided by the specific needs of youth with OCD and their families (e.g., accommodation, conflict). The first phase of the proposed study will involve an open case series in order to assess the utility of the PFIT protocol and feasibility of training other therapists and using the manual with a range of patient presentations. The second phase will involve a small controlled feasibility trial evaluating the extent to which recruitment, randomization, and implementation of the control condition are viable for further study. It is hypothesized that the PFIT treatment will be feasible to implement and will yield higher levels of patient satisfaction compared to treatment as usual.

DETAILED DESCRIPTION:
Pediatric Obsessive Compulsive Disorder (OCD) is among the most common disorders of childhood, affecting between 1 and 3% of the youth population. The disorder is associated with substantial impairment in academic, social, and family functioning, and it carries a host of risks as youth age into adulthood. Cognitive behavioral therapy (CBT) has emerged as the treatment of choice for pediatric OCD, with typical treatment protocols involving exposure to feared stimuli, identification and evaluation of maladaptive beliefs, relaxation training, and behavioral rewards. Although these techniques have produced favorable results, one third of youth with OCD do not demonstrate significant response to treatment and many of those who do respond continue to evidence some degree of symptoms and impairment.

Efforts to improve therapy outcomes for youth with OCD increasingly have attempted to augment individual CBT with greater family involvement. These programs typically involve psychoeducation about OCD as well as general behavioral strategies for enhancing adherence to treatment. Although current family-focused treatments vary with regard to the nature and extent of parent involvement, to date, the incremental benefit of adding a family treatment component to traditional individual treatment remains unclear. Indeed, there does not appear to be a relation between the degree of family involvement and degree of treatment response, and current family treatments do not appear to affect change in family beliefs or behaviors.

This picture suggests that either family involvement does not contribute to significant improvement in child outcomes or that current treatments may not be sufficiently focused on features of the home environment that are relevant for shaping and maintaining OCD symptoms. Building from theoretical literature which identifies familial blame and accommodation as key characteristics that are important for course and outcome in OCD, we have developed a novel family intervention for use in treating pediatric OCD. Using techniques that are well established, Positive-Family Interaction Therapy (P-FIT) attempts to reduce family blame, accommodation, and conflict and to enhance family cohesion in high stress, high conflict families.

The goals of this study are to investigate a manualized P-FIT program for youth with OCD first with a small open trial of up to ten families to investigate the feasibility and tolerability of the treatment and then with a randomized trial (the main study) to assess its incremental efficacy over usual care (i.e., individual cognitive behavioral therapy). For the initial pilot stage, up to four children between the ages of 9-17 will be treated with P-FIT through the UCLA Child OCD, Anxiety, and Tic Disorders Program after completing a diagnostic evaluation to confirm eligibility. During this pilot study, procedures and materials for the manual will be refined and finalized for the controlled trial. The treatment will consist of 12 sessions of standard cognitive behavioral therapy that is augmented with a novel 6-session family focused treatment module. Assessments involving interviews, questionnaires, and several short tasks will be conducted at the beginning, midpoint and end of the treatment. We will also follow up with families 3 months following treatment in order to assess durability of any treatment gains. Study staff will meet weekly to discuss each open trial therapy session, including the feasibility, efficacy, and acceptability of the treatment manual, and make adjustments as needed. Once this group reaches consensus regarding the suitability of the manual, recruitment into the open trial will end and subsequent eligible families will be invited to participate in the randomized controlled trial (the main study).

Over the course of the main study, 40 youngsters will be randomized to receive either individual child-centered cognitive behavioral therapy (ICBT) or the P-FIT intervention (ICBT + 6 sessions of family treatment). All subjects regardless of response status will be evaluated at all scheduled assessment points. In addition to comprehensive parent, child, and clinician reports, the primary outcome variables will be assessed by blind independent evaluators. Manualized intervention and assessment protocols plus state-of-the art quality assurance (i.e., weekly supervision with an expert clinician specializing specifically in OCD treatment) and adverse event monitoring procedures will insure participant safety. Results from this investigation will be used to support a larger controlled comparative trial comparing the degree to which P-FIT improves outcomes for youth with OCD above and beyond current available treatments.

ELIGIBILITY:
Inclusion Criteria:

* Ages 9 to 17 years old, inclusive, at the point of consent.
* DSM-IV criteria for a primary diagnosis of OCD on the Anxiety Disorders Interview Schedule for DSM-IV (Silverman & Albano, 1996).
* CYBOCS >15
* Impaired family functioning as indicated by unhealthy FES conflict or PABS Blame scores (based on published FES clinic norms and distribution of PABS scores from our clinic population)
* Availability of primary caregivers to participate in the family-treatment module
* Informed parental consent and child assent.

Exclusion Criteria:

* Participants with the following DSM-IV psychiatric disorders will be excluded: Bipolar disorder, PTSD, substance abuse/dependence, conduct disorder, PDD, schizophrenia, or mental retardation. Youth with other comorbid disorders (e.g., anxiety, ADHD, ODD, TS) will be eligible as long as these disorders are secondary to OCD in terms of severity and impairment and do not require immediate initiation of treatment.
* Recent treatment with psychotropic medication within 6 weeks of study entry for fluoxetine, within 2 weeks for other SSRIs, and 4 weeks for neuroleptics.
* Child has failed a previous trial of CBT for anxiety within the previous 2 years judged adequate by at least 10 treatment sessions over a period of less than 1 year.
* Child has a major neurological disorder or a major medical illness that would interfere with participation in the study (e.g., frequent hospitalizations, frequent school absences).
* Child poses a significant risk for dangerousness to self or to others that makes participating inadvisable.
* Child and/or parent is non-English speaking (unable to complete measures, IE ratings, or treatment without the assistance of a dedicated translator).
* Parents will be excluded based on the following criteria: (a) apparent parental psychiatric disturbance of sufficient severity to contraindicate study participation and/or (b) insufficient command of the English language. Parent psychiatric status will be screened using the Brief Symptom Inventory (BSI). This process will include review of available study assessment measures and further interview with the parent, if needed. Dr. Peris or another senior licensed clinician will meet with all parents deemed ineligible for study participation based on their psychiatric status to inform them of study ineligibility and reasons for exclusion and to provide at least two referrals will be provided for further care.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
OCD symptom severity on the Children's Yale Brown Obsessive Compulsive Scale (CYBOCS) | Post-treatment (week 12)
  Treatment outcome will be evaluated based on decreases in total OCD symptom severity as measured by the CYBOCS.

CONTACTS AND LOCATIONS:
Overall Officials: Tara S Peris, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Derived] Peris TS, Rozenman MS, Sugar CA, McCracken JT, Piacentini J. Targeted Family Intervention for Complex Cases of Pediatric Obsessive-Compulsive Disorder: A Randomized Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2017 Dec;56(12):1034-1042.e1. doi: 10.1016/j.jaac.2017.10.008. Epub 2017 Oct 14. PMID 29173737